CLINICAL TRIAL: NCT06173843
Title: Effect of Occupational Exposures on Cancer Pathophysiology Among Firefighters
Brief Title: Occupational Exposures Among Firefighters
Status: Recruiting | Type: Observational
Sponsor: Vincere Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: VCC-PFAS-001
Record Dates: First submitted 2023-12-07; First posted 2023-12-18 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Cancer
Keywords: Cancer; Occupational exposure
MeSH Terms: conditions — Neoplasms | interventions — phosphoribosylformylglycinamidine synthetase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Firefighters
  Interventions: Other: PFAS / heavy metal testing, exposures
- Non-Firefighters
  Interventions: Other: PFAS / heavy metal testing, exposures

INTERVENTIONS:
Other: PFAS / heavy metal testing, exposures — PFAS / heavy metal concentrations, exposure survey

SUMMARY:
This study aims to understand the effect of occupational exposures, including PFAS exposures, among firefighters.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older; any gender
* Currently (or previously) employed as a firefighter, full-time or part-time, participating in Vincere's First Responder Cancer Screening Program
* Willing to provide a blood, urine, and/or tissue sample
* Able to provide informed consent to participate in the study

(A small group of non-firefighters will be enrolled to act as a comparison group)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Actively working or retired firefighters of any adult age, any gender and any demographic group are eligible, with no limitations regarding general health status other than those specified in the protocol Eligibility Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Exposures associated with elevated PFAS | 5 years

SECONDARY OUTCOMES:
Cancer rates | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Vincere Cancer Center, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No